CLINICAL TRIAL: NCT01889121
Title: Retrospective Analysis of the Utility Formal Psychosocial Support in Enhancing the Outcome of Pregnancies in Opiate-addicted Pregnant Women in Agonist Maintenance Programs
Brief Title: Utility of Psychosocial Intervention in Improving Outcome for Methadone-exposed Infants and Their Mothers
Acronym: HOPE
Status: Completed | Type: Observational
Sponsor: Dr. Henry Akinbi (Other)
Responsible Party: Sponsor-Investigator, Dr. Henry Akinbi, Associate Professor, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Other Study IDs: HOPE_Methadone
Record Dates: First submitted 2013-06-24; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Methadone maintenance program: Mothers on methadone treatment at time of delivery who delivered at Good Samaritan Hospital but were not enrolled in psychosocial intervention offered through the HOPE (Helping Opiate-addicted Pregnant women Evolve) program.
- Psychosocial intervention: Pregnant women who were in methadone maintenance program PLUS structured psychosocial intervention at the time of delivery (HOPE Program).
  Interventions: Behavioral: Structured psychosocial intervention

INTERVENTIONS:
Behavioral: Structured psychosocial intervention — This is retrospective analysis of two groups of opiate-addicted pregnant women: 1) Pregnant women in methadone maintenance program 2) Pregnant women in methadone maintenance program AND structured psychosocial intervention
  Groups: Psychosocial intervention

SUMMARY:
Opiate drug abuse/addiction is a significant co-morbidity in pregnancy. Opiate maintenance program enhances the outcome of pregnancies for the mother and the infant. Our objective was to assess if provision of structured psychosocial support in addition to methadone maintenance program adds incremental benefits with regards to the outcome of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Positive Methadone tox screen
* Received care at Good Samaritan Hospital in Cincinnati
* Delivered at Good Samaritan Hospital

Exclusion Criteria:

* Twin gestation
* Sever congenital anomalies
* Conditions requiring transfer to quaternary hospital

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Opiate abusing pregnant women who received their prenatal care through Good Samaritan Faculty Medical Center and were getting methadone maintenance therapy
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Percentage of newborns in each group that required pharmacological treatment for neonatal abstinence syndrome | Birth until discharge
  Infants delivered to mothers that are maintained on methadone are at risk for neonatal abstinence syndrome. Psychosocial support is provided to pregnant women in methadone maintenance program to impact the outcome of the infants. The percentage of infants requiring pharmacotherapy would be expected to be reduced by the addition of psychosocial intervention to methadone maintenance program.

SECONDARY OUTCOMES:
Gestational age at which the infants were delivered. | Gestational age at delivery.
  Addiction of pregnant women to opiate drugs is associated with preterm delivery. The gestational ages of infants delivered to women in the two groups will be compared for statistically significant differences.
Percentage of infants that are small for gestational age. | Gestional period.
  Addiction to opiates is associated with fetal growth restriction. This study compared the proportion of infants who are <90th percentile for gestational age in both groups.
Anthropometric measurements at birth | Measurements at birth.
  Differences between the mean birth weight, Length and head circumference at birth were compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States